CLINICAL TRIAL: NCT07248891
Title: Comprehensive Study of Associated Factors With Type 2 Diabetes in Mexico: Protocol
Brief Title: Type 2 Diabetes and Associated Factors in Mexico
Status: Enrolling by invitation | Type: Observational
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2024-785-007
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Kidney Disease; Diabetic Nephropathy
Keywords: Glycemic Control; Glycated Hemoglobin; Genes; Transcriptome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood samples were collected for serum and RNA. A 6 mL vacutainer tube was centrifuged to obtain serum for biochemical analysis and complete blood count. RNA was isolated from blood using standard extraction kits for transcriptomic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Type 2 Diabetes: This cohort included adult patients (≥18 years) with a confirmed diagnosis of Type 2 Diabetes Mellitus. Participants were recruited from Family Medicine Units in Coahuila, Jalisco, and Veracruz, Mexico. All underwent clinical evaluation, lifestyle and dietary assessments, functional testing, and blood sampling for biochemical and transcriptomic analysis
  Interventions: Other: Clinical and Molecular Assessment

INTERVENTIONS:
Other: Clinical and Molecular Assessment — Participants underwent clinical examination, lifestyle and dietary questionnaires, functional testing (six-minute walk test), and blood sampling for biochemical and transcriptomic analysis.

SUMMARY:
The goal of this observational cross-sectional multicenter study is to identify clinical, lifestyle, metabolic, inflammatory, and genetic factors associated with glycemic control and complications of Type 2 Diabetes (T2D) in adult patients in Mexico.

The main questions it aims to answer are:

Which molecular and clinical factors are associated with poor glycemic control (HbA1c > 7%)?

Which factors are linked to the presence of diabetic nephropathy (GFR < 60 mL/min/1.73 m²)?

Participants:

Provide informed consent and clinical history.

Undergo a clinical and physical evaluation (including six-minute walk test).

Complete lifestyle, dietary, and therapeutic adherence questionnaires.

Provide blood samples for biochemical, inflammatory, and transcriptomic (RNA-Seq) analysis.

Researchers integrate clinical, biochemical, and transcriptomic data using statistical modeling to identify a characteristic molecular fingerprint of poor metabolic control and diabetes-related complications.

DETAILED DESCRIPTION:
This observational, cross-sectional, multicenter study evaluates adult patients with Type 2 Diabetes (T2D) in three regions of Mexico (Coahuila, Jalisco, and Veracruz) to explore the interaction of clinical, lifestyle, metabolic, inflammatory, and genetic factors with glycemic control and diabetes-related complications. A total of 1,000 participants are recruited from Family Medicine Units, where they undergo standardized clinical assessments, lifestyle and dietary evaluations, functional testing, and laboratory investigations.

Blood samples are collected for biochemical parameters, inflammatory markers, and transcriptomic (RNA-Seq) analysis. Glycemic control is assessed through HbA1c, while diabetic nephropathy is determined using estimated glomerular filtration rate (eGFR). Multivariate and principal component analyses are applied to integrate clinical, biochemical, and molecular information.

The study aims to identify a pathological molecular fingerprint that characterizes poor metabolic control and diabetic complications. By combining clinical and molecular profiles, this protocol seeks to contribute evidence for improving risk stratification, clinical decision-making, and future public health strategies targeting T2D in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Established diagnosis of Type 2 Diabetes Mellitus (T2D).
* Patients receiving care at Family Medicine Units in Coahuila, Jalisco, or Veracruz.
* Willingness to voluntarily participate in the study.
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Pregnant or lactating mother
* Current use of steroids
* Concomitant illness with inflammatory or autoimmune component (rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, psoriatic arthritis, gout).
* Tobacco use (in the last 3 months).
* History of cerebrovascular disease, heart failure or kidney failure that required hospitalization in the previous month.
* History of infection in the previous 10 days (respiratory tract infection, gastroenteritis, urinary tract infection, soft tissue infection).
* Severe obesity with BMI > 40 kg/m2. History of bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Type 2 Diabetes Mellitus are recruited from three Family Medicine Units of the Mexican Social Security Institute (IMSS): FMU No. 10 in Coahuila, FMU No. 181 in Jalisco, and FMU No. 30 in Veracruz. The study population represents individuals receiving primary care for diabetes management in different regions of Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (% HbA1c) | At baseline (single cross-sectional assessment).
  Proportion of participants with poor glycemic control, defined as HbA1c > 7%.
Diabetic Nephropathy (eGFR) | At baseline (single cross-sectional assessment).
  Presence of diabetic nephropathy defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m².

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Ferreira Hermosillo, Researcher, Study Director — Medical Research Unit in Endocrine Diseases
Locations (3):
- Mexico (3):
  - Coordinación de Investigación en Salud, Mexico City, Mexico City
  - División de Investigación en Salud, Mexico City, Mexico City
  - Instituto Mexicano del Seguro Social, Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: Undecided
At this time, the plan to share individual participant data (IPD) is undecided. The investigators are considering whether de-identified clinical and molecular data can be shared with other researchers while ensuring compliance with IMSS institutional policies, national regulations, and participant privacy protection.

REFERENCES:
- [Background] Francisco V, Pino J, Gonzalez-Gay MA, Mera A, Lago F, Gomez R, Mobasheri A, Gualillo O. Adipokines and inflammation: is it a question of weight? Br J Pharmacol. 2018 May;175(10):1569-1579. doi: 10.1111/bph.14181. Epub 2018 Apr 10. PMID 29486050
- [Result] Basto-Abreu A, Lopez-Olmedo N, Rojas-Martinez R, Aguilar-Salinas CA, Moreno-Banda GL, Carnalla M, Rivera JA, Romero-Martinez M, Barquera S, Barrientos-Gutierrez T. Prevalencia de prediabetes y diabetes en Mexico: Ensanut 2022. Salud Publica Mex. 2023 Jun 13;65:s163-s168. doi: 10.21149/14832. Spanish. PMID 38060942
- [Result] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- See also: Revista Médica del Instituto Mexicano del Seguro Social — https://revistamedica.imss.gob.mx/index.php/revista_medica/article/view/6386/5673